CLINICAL TRIAL: NCT06380530
Title: Advanced Surgical Simulation Processes in the Correction of Skeletal Defects and Deformities
Acronym: SIMULA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Collaborators: Ospedale Pediatrico Bambino Gesù (Unknown); Istituto Giannina Gaslini (Other); Galeazzi Orthopedic Institute (Unknown); Istituto Nazionale Tumori Regina Elena (Unknown); Policlinico San Matteo (Unknown); Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SIMULA
Record Dates: First submitted 2024-04-18; First posted 2024-04-24 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Musculoskeletal Deformity; Musculoskeletal Abnormalities; Musculoskeletal Disorder
Keywords: Virtual Surgical Planning; Patient-Specific instrument; Graft-Specific instrument; Pediatric Orthopedics
MeSH Terms: conditions — Musculoskeletal Abnormalities; Musculoskeletal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pediatric patients with musculoskeletal diseases (Experimental): Children, adolescents, and young adults suffering from musculoskeletal disorders (MMD) who exhibit complex conditions characterized by rare and severe anomalies in skeletal development. These abnormalities may affect bones, joints, and musculotendinous structures.
  Interventions: Procedure: Deformity correction

INTERVENTIONS:
Procedure: Deformity correction — Surgeries to correct bone defomity, supported by the use of preoperative planning and/or patient-specific instruments

SUMMARY:
Virtual Surgical Planning (VSP), Computer-Aided Surgical Simulation (CASS) for bone corrections, and the customization of implants and devices through 3D printing, known as Patient-Specific Instruments (PSI) and Graft-Specific Instruments (GSI), are assuming increasingly central roles in orthopedic clinical and surgical practice.

One area witnessing notable advancement is the treatment of musculoskeletal disorders (MMS) in children, adolescents, and young adults. These disorders involve severe and rare abnormalities in skeletal formation and development across three-dimensional planes, often affecting multiple limbs. Managing such deformities is complex, challenging to standardize, and prone to unpredictable clinical, radiographic, and functional outcomes.

The application of 3D modeling and printing technologies offers a deeper understanding of deformities and facilitates improved prediction, precision, reproducibility, and safety in surgical interventions.

The Musculoskeletal Apparatus Network (RAMS Network) centers are equipped with advanced 3D laboratories for surgical simulation and planning, aligned with the overarching goal of improving surgery quality through "in-silico" medicine (ISM) principles.

At present, numerous complex surgeries involving Virtual Surgical Planning (VSP) and sterilizable 3D-printed Patient-Specific Instruments (PSI) and/or Graft-Specific Instruments (GSI) are being simulated and performed at the Rizzoli Institute. Preliminary data from previous protocols indicate a significant reduction in surgical time with the implementation of VSP and the utilization of PSI and GSI.

The aim of this study is to enhance the current process of simulating, planning, and designing surgical support tools within 3D Printing Point-of-Care (3D POC) facilities. To achieve this, it is imperative to expand case volumes and systematically organize, categorize, and standardize simulation and planning procedures.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of musculoskeletal disease (MSD) of the limbs;
* Need for mono- or polyaxial correction by one or more osteotomies;
* Presence of specific consent to participate in the trial;

Exclusion Criteria:

* Patients who refuse to participate in the study
* Patients who do not undergo radiological follow-up examinations for VSP or for whom the radiological record is insufficient to conduct VSP;
* Patients who undergo different interventions for correction of MSD (growth modulation interventions by epiphysiodesis and hemiepiphysiodesis, progressive correction by external circular/hexapodal fixation);
* Pregnant or lactating women

Ages: 2 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-10-31 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Achieved skeletal corrections | At baseline (day 0)
  Assessment of achieved skeletal corrections compared to planned corrections, measured on standard radiographs or CT scans depending on the type of deformity corrected
Achieved skeletal corrections | After 1 year
  Assessment of achieved skeletal corrections compared to planned corrections, measured on standard radiographs or CT scans depending on the type of deformity corrected

SECONDARY OUTCOMES:
Operating room times | At baseline (day 0)
  Operating room times for each planned procedure
Fluoroscopy times | At baseline (day 0)
  Fluoroscopy times for each planned procedure
Blood loss | At baseline (day 0)
  Blood loss for each patient
Intra- and peri-operative complications | At baseline (day 0)
  Intra- and peri-operative complications for each patient
Suitability of PSIs | At baseline (day 0)
  Suitability of PSIs in relation to the planned surgery
Suitability of GSIs | At baseline (day 0)
  Suitability of GSIs, if needed, in relation to the planned surgery
Suitability of bone graft | At baseline (day 0)
  Suitability of bone graft, if needed, in relation to the planned surgery
Clinical-functional outcome | At baseline (day 0)
  Clinical-functional outcome will be assessed by preoperative and one-year follow-up administration of the Pediatric Outcome Data Collection Instrument (PODCI) questionnaire for pediatric patients or the Short Form Health Survey 36 (SF-36) for young adults
Clinical-functional outcome | After 1 year
  Clinical-functional outcome will be assessed by preoperative and one-year follow-up administration of the Pediatric Outcome Data Collection Instrument (PODCI) questionnaire for pediatric patients or the Short Form Health Survey 36 (SF-36) for young adults

OTHER OUTCOMES:
Cost analysis | At baseline (day 0)
  The cost analysis will entail evaluating expenses associated with various components, including imaging required for planning, production of 3D-printed instrumentation such as PSIs and GSIs, and bone grafts. Additionally, human costs for planning will be considered. Surgical-related costs will be assessed by comparing them with those of traditional surgeries to gauge the cost-effectiveness of the procedure, taking into account the achieved correction and the necessity for additional procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Pierfrancesco Costici, MD, Principal Investigator — Ospedale Pediatrico Bambin Gesù; Giorgio Marrè Brunenghi, MD, Principal Investigator — Istituto Giannina Gaslini; Fabio Verdoni, MD, Principal Investigator — Galeazzi Orthopedic Institute; Roberto Biagini, MD, Principal Investigator — Istituto Nazionale Tumori Regina Elena; Gianluigi Pasta, MD, Principal Investigator — Policlinico San Matteo; Tommaso Bonanzinga, MD, Principal Investigator — Istituto Clinico Humanitas
Locations (7):
- Italy (7):
  - IRCCS Istituto Ortopedico Rizzoli, Bologna, BO
  - Istituto Clinico Humanitas, Rozzano, MI
  - Istituto Giannina Gaslini, Genova
  - Galeazzi Orthopedic Institute, Milan
  - Policlinico San Matteo, Pavia
  - Istituto Nazionale Tumori Regina Elena, Roma
  - Ospedale Pediatrico Bambino Gesù, Roma

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] R. Michaels et al., "3D printing in surgical simulation: emphasized importance in the COVID-19 pandemic era," https://doi.org/10.2217/3dp-2021-0009, vol. 5, no. 1, pp. 5-9, May 2021, doi: 10.2217/3DP-2021-0009.
- [Background] S. Dash, S. K. Shakyawar, M. Sharma, and S. Kaushik, "Big data in healthcare: management, analysis and future prospects," J Big Data, vol. 6, no. 1, pp. 1-25, Dec. 2019, doi: 10.1186/S40537-019-0217-0/FIGURES/6.
- [Background] G. Pravettoni and S. Triberti, "A 'P5' Approach to Healthcare and Health Technology," P5 eHealth: An Agenda for the Health Technologies of the Future, pp. 3-17, 2020, doi: 10.1007/978-3-030-27994-3_1.
- [Background] Anaya JM, Duarte-Rey C, Sarmiento-Monroy JC, Bardey D, Castiblanco J, Rojas-Villarraga A. Personalized medicine. Closing the gap between knowledge and clinical practice. Autoimmun Rev. 2016 Aug;15(8):833-42. doi: 10.1016/j.autrev.2016.06.005. Epub 2016 Jun 11. PMID 27302209
- [Background] Coppola L, Cianflone A, Grimaldi AM, Incoronato M, Bevilacqua P, Messina F, Baselice S, Soricelli A, Mirabelli P, Salvatore M. Biobanking in health care: evolution and future directions. J Transl Med. 2019 May 22;17(1):172. doi: 10.1186/s12967-019-1922-3. PMID 31118074
- [Background] Pop B, Fetica B, Blaga ML, Trifa AP, Achimas-Cadariu P, Vlad CI, Achimas-Cadariu A. The role of medical registries, potential applications and limitations. Med Pharm Rep. 2019 Jan;92(1):7-14. doi: 10.15386/cjmed-1015. Epub 2019 Jan 15. PMID 30957080
- [Background] Dorsey ER. The new platforms of health care. NPJ Digit Med. 2021 Jul 15;4(1):112. doi: 10.1038/s41746-021-00478-5. PMID 34267312
- [Background] Tumiene B, Graessner H, Mathijssen IM, Pereira AM, Schaefer F, Scarpa M, Blay JY, Dollfus H, Hoogerbrugge N. European Reference Networks: challenges and opportunities. J Community Genet. 2021 Apr;12(2):217-229. doi: 10.1007/s12687-021-00521-8. Epub 2021 Mar 17. PMID 33733400
- [Background] Vivarelli L, Govoni M, Attala D, Zoccali C, Biagini R, Dallari D. Custom Massive Allograft in a Case of Pelvic Bone Tumour: Simulation of Processing with Computerised Numerical Control vs. Robotic Machining. J Clin Med. 2022 May 15;11(10):2781. doi: 10.3390/jcm11102781. PMID 35628908
- [Background] Benedetti MG, et al. Prot. CHILD-DEROT. 'Studio pilota per la pianificazione del trattamento alterazioni torsionali dell'arto inferiore nei bambini affetti da paralisi cerebrale infantile mediante valutazione integrata morfologica e funzionale.' CE AVEC 718/2021/Oss/IOR. 30/09/2021.
- [Background] L. Frizziero et al., "Computer-aided surgical simulation for correcting complex limb deformities in children," Applied Sciences (Switzerland), vol. 10, no. 15, Aug. 2020, doi: 10.3390/app10155181.
- [Background] Raza M, Murphy D, Gelfer Y. The effect of three-dimensional (3D) printing on quantitative and qualitative outcomes in paediatric orthopaedic osteotomies: a systematic review. EFORT Open Rev. 2021 Feb 1;6(2):130-138. doi: 10.1302/2058-5241.6.200092. eCollection 2021 Feb. PMID 33828856
- [Background] Grassi FR, Grassi R, Vivarelli L, Dallari D, Govoni M, Nardi GM, Kalemaj Z, Ballini A. Design Techniques to Optimize the Scaffold Performance: Freeze-dried Bone Custom-made Allografts for Maxillary Alveolar Horizontal Ridge Augmentation. Materials (Basel). 2020 Mar 19;13(6):1393. doi: 10.3390/ma13061393. PMID 32204393
- [Background] Frizziero L, Santi GM, Leon-Cardenas C, Donnici G, Liverani A, Papaleo P, Napolitano F, Pagliari C, Di Gennaro GL, Stallone S, Stilli S, Trisolino G, Zarantonello P. In-House, Fast FDM Prototyping of a Custom Cutting Guide for a Lower-Risk Pediatric Femoral Osteotomy. Bioengineering (Basel). 2021 May 26;8(6):71. doi: 10.3390/bioengineering8060071. PMID 34073324
- [Background] L. Frizziero et al., "Paediatric orthopaedic surgery with 3D printing: Improvements and cost reduction," Symmetry (Basel), vol. 11, no. 10, Oct. 2019, doi: 10.3390/sym11101317.
- [Background] L. Frizziero et al., "An innovative and cost-advantage cad solution for cubitus varus surgical planning in children," Applied Sciences (Switzerland), vol. 11, no. 9, May 2021, doi: 10.3390/app11094057.
- [Background] "3D-MALF: 'Modelli 3D-printing nel planning preoperatorio del paziente pediatrico affetto da malformazioni congenite. Studio pilota.' - CE AVEC: 356/2018/Sper/IOR".
- [Background] "3D-MALF II: 'Innesti ossei personalizzati mediante analisi tridimensionale nelle deformità scheletriche in età pediatrica' - CE AVEC: 301/2022/Sper/IOR."
- [Background] L. Frizziero et al., "New Methodology for Diagnosis of Orthopedic Diseases through Additive Manufacturing Models," Symmetry 2019, Vol. 11, Page 542, vol. 11, no. 4, p. 542, Apr. 2019, doi: 10.3390/SYM11040542.
- [Background] L. Frizziero et al., "Effectiveness assessment of CAD simulation in complex orthopedic surgery practices," Symmetry (Basel), vol. 13, no. 5, May 2021, doi: 10.3390/sym13050850.
- [Background] F. Osti et al., "CT conversion workflow for intraoperative usage of bony models: From DICOM data to 3D printed models," Applied Sciences (Switzerland), vol. 9, no. 4, Feb. 2019, doi: 10.3390/app9040708.
- [Background] G. Durastanti, C. Belvedere, M. Ruggeri, D. M. Donati, B. Spazzoli, and A. Leardini, "A Pelvic Reconstruction Procedure for Custom-Made Prosthesis Design of Bone Tumor Surgical Treatments," Applied Sciences 2022, Vol. 12, Page 1654, vol. 12, no. 3, p. 1654, Feb. 2022, doi: 10.3390/APP12031654.
- [Background] Alessandri G, Frizziero L, Santi GM, Liverani A, Dallari D, Vivarelli L, Di Gennaro GL, Antonioli D, Menozzi GC, Depaoli A, Rocca G, Trisolino G. Virtual Surgical Planning, 3D-Printing and Customized Bone Allograft for Acute Correction of Severe Genu Varum in Children. J Pers Med. 2022 Dec 12;12(12):2051. doi: 10.3390/jpm12122051. PMID 36556271
- [Background] Archunan MW, Petronis S. Bone Grafts in Trauma and Orthopaedics. Cureus. 2021 Sep 4;13(9):e17705. doi: 10.7759/cureus.17705. eCollection 2021 Sep. PMID 34650879
- [Background] Depaoli A, Menozzi GC, Di Gennaro GL, Ramella M, Alessandri G, Frizziero L, Liverani A, Martinelli D, Rocca G, Trisolino G. The Flipping-Wedge Osteotomy: How 3D Virtual Surgical Planning (VSP) Suggested a Simple and Promising Type of Osteotomy in Pediatric Post-Traumatic Forearm Deformity. J Pers Med. 2023 Mar 19;13(3):549. doi: 10.3390/jpm13030549. PMID 36983730
- [Background] Customized Bone Allografts by 3D-printing - Full Text View - ClinicalTrials.gov." https://classic.clinicaltrials.gov/ct2/show/NCT05700526?term=malf&cntry=IT&draw=2&rank=1 (accessed Aug. 21, 2023)
- [Background] Frizziero L, Santi GM, Leon-Cardenas C, Ferretti P, Sali M, Gianese F, Crescentini N, Donnici G, Liverani A, Trisolino G, Zarantonello P, Stallone S, Di Gennaro GL. Heat Sterilization Effects on Polymeric, FDM-Optimized Orthopedic Cutting Guide for Surgical Procedures. J Funct Biomater. 2021 Nov 19;12(4):63. doi: 10.3390/jfb12040063. PMID 34842761
- See also: Customized Bone Allografts by 3D-printing (3D-MALF 2 protocol) — https://classic.clinicaltrials.gov/ct2/show/NCT05700526?term=malf&cntry=IT&draw=2&rank=1